CLINICAL TRIAL: NCT02147106
Title: Use of Video Consultation in Follow-up Care for Patients With a NeuroEndocrine Tumor: a Feasibility Study (VIDEO-NET Study)
Brief Title: Use of Video Consultation in Follow-up Care for Patients With a Neuroendocrine Tumor: a Feasibility Study
Acronym: VIDEO-NET
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: VIDEO-NET-2014
Record Dates: First submitted 2014-05-19; First posted 2014-05-26 (Estimated); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Neuroendocrine Tumor
Keywords: Neuroendocrine tumor; Videoconsultation; Feasibility
MeSH Terms: conditions — Neuroendocrine Tumors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Videoconsultation: Performing two videoconsulations with the treating medical oncologist
  Interventions: Other: Videoconsultation

INTERVENTIONS:
Other: Videoconsultation

SUMMARY:
Rationale: Patients with neuroendocrine tumors (NET) have a rare disease. Due to treating patients with a neuroendocrine tumor in 'NET knowledge centers' patients often have to travel long distances for follow-up visits at the outpatient clinic. Patients whose medical condition allows videoconsultation could save time by replacing outpatient clinic visits through videoconsultation for receiving follow-up care. Therefore, in this study we aim to introduce videoconsultation as a alternative for follow-up outpatient clinic visits in NET patients.

Objective: The primary objective is to assess if use of videoconsultation in follow-up care for NET patients is feasible. We hypothesize that videoconsultation is a suitable medium for providing follow-up care in NET patients. Secondary objectives are to explore the amount of time videoconsultation takes in comparison with outpatient clinic visits and the acceptability and satisfaction of physicians and patients with using videoconsultation in follow-up care.

Study design: The present study is a single-centre prospective feasibility study.

Study population: Adult NET patients under surveillance or treatment of the department Medical Oncology at the University Medical Centre Groningen (UMCG) whose medical condition allows videoconsultation will be invited to participate.

Intervention: Patient who give informed consent will participate in the study. Participants will receive follow-up care through videoconsultation instead of conventional visits at the outpatient clinic.

Main study parameters/endpoints: The main endpoint is the feasibility of videoconsultation for follow-up care in NET patients. We hypothesize that videoconsultation is a suitable medium for providing follow-up care.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age ≥ 18 yrs
* Grade I or II (low and intermediate grade) NET with any primary tumor type or disease stage
* Have access to required equipment/technology for performing videoconsultation

Exclusion Criteria:

* Newly referred NET patients, who are visiting the department of Medical Oncology at the UMCG for the first time
* Recently diagnosed NET patients, who are in the diagnostic phase of the disease
* NET patients who frequently require blood tests, consultation or physical examination
* A hearing or visual impairment, which would make videoconsultation difficult

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Neuroendocrine tumor patients (grade 1 and 2) whose medical condition allows videoconsultation.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2014-05; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Feasibility | 1 year
  Participation rates, reason for declining participation, number of completed videoconsultations, dropout rate and reason for dropout will be noted in study records to evaluate feasibility of videoconsultation

SECONDARY OUTCOMES:
Amount of time | 1 year
  The amount of time NET patients are spending with videoconsultation in comparison with conventional outpatient clinic visits.
Acceptability and satisfaction of patients | 1 year
  The acceptability and satisfaction of patients with the use of videoconsultation will be assessed with a questionnaire and open-ended questions.
Acceptability and satisfaction of physicians | 1 year
  The acceptability and satisfaction of physicians with the use of videoconsultation will be assessed with a questionnaire and open-ended questions.

CONTACTS AND LOCATIONS:
Overall Officials: A.M.E. Walenkamp, MD PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands